CLINICAL TRIAL: NCT01778998
Title: Impact of Incision Size and Architecture on Wound Stability and Astigmatism in Cataract Surgery: an Exploratory Study
Acronym: INCISIONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Univ.-Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: INCISIONS
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Cataract
Keywords: incision; pre-cut; wound architecture; OCT
MeSH Terms: conditions — Cataract; Surgical Wound

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MICS-group (Active Comparator)
  Interventions: Procedure: MICS-group
- SICS-group (Active Comparator)
  Interventions: Procedure: SICS-group
- SICS pre-cut (Active Comparator)
  Interventions: Procedure: SICS pre-cut
- SICS stab-incision (Active Comparator)
  Interventions: Procedure: SICS stab-incision

INTERVENTIONS:
Procedure: MICS-group — Micro incision cataract surgery is done
  Arms: MICS-group
Procedure: SICS-group — small incision cataract surgery is done
  Arms: SICS-group
Procedure: SICS pre-cut — Small incision cataract surgery with pre-cut is done
  Arms: SICS pre-cut
Procedure: SICS stab-incision — Small incision cataract surgery with stab-incision is done
  Arms: SICS stab-incision

SUMMARY:
One of the most recent advances in cataract surgery is microincisional phacoemulsification (MICS). Through small incisions of 2.0 mm and less the lens material is emulsified either bimanually or with a thin single coaxial hand-piece. The possible advantages are lower induced corneal astigmatism1, 2, possibly a lower incidence of infection due to higher resistance of the wound to deformation3 and a lower risk of complications such as iris prolapse during surgery in patients at risk such as with intraoperative floppy iris syndrome (IFIS). Additional factors that have to be taken into account are the construction and the position of the incision and the influence of the extraocular force on the wound morphology.4 Another effect that may influence the wound architecture is stromal hydration at the end of surgery.5 Wound architecture has recently been assessed6-9 using optical coherence tomography. Elkady et al.10 observed the wound architecture in MICS cases focusing on corneal thickness and the incision angle. However, none of these studies observed the effect of the wound architecture on post-operative astigmatism. Furthermore, all observations in the past have been performed in the post-operative period only and information concerning the wound architecture intra-operatively is missing. A recently launched CE-marked intra-operative OCT allows observing the wound architecture intra-operatively.

One aim of the study is to assess the influence of the intra-operative wound architecture using a similar grading system as used by Calladine and Packard (2007)7 on the resistance to deformation of the wound and the surgically induced astigmatism in MICS and small incision cataract surgery (SICS). In a second part of this exploratory study the effect of a hinged incision with a pre-cut should be assessed along the same line

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Any ophthalmic abnormality that could compromise the measurements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
o Correlation between a wound architecture score (developed during the study) and the post-operative astigmatism for the "MICS", the "SICS", the "SICS pre-cut" and the "SICS stab-incision" group | pre-operatively to one day post-operativly

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — VIROS - Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Vienna, Austria